CLINICAL TRIAL: NCT00819767
Title: An Eight-week, Randomized, Double-blind, Parallel-group, Pilot Study to Evaluate the Efficacy and Safety of Aliskiren 300 mg in Comparison With Valsartan 320 mg in Patients With Mild to Moderate Hypertension During Exercise After a Missed Dose
Brief Title: Efficacy and Safety of Aliskiren in Patients With Mild to Moderate Hypertension During Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2406
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: hypertension; systolic blood pressure; exercise test; cardiovascular disease; aliskiren; valsartan
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — aliskiren; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental): For the first week of the 8 week treatment period, patients received aliskiren 150 mg, placebo to aliskiren, and 2 capsules of placebo to valsartan. For the remaining 7 weeks of the study, patients received aliskiren 300 mg (two 150 mg tablets) and 2 capsules of placebo to valsartan. The tablets and capsules (2 of each) were taken orally once daily each morning. To evaluate a missed dose, the last dose of medication was administered at the clinic, and the patient was scheduled to return 2 days later for exercise testing (8 weeks + 2 days).
  Interventions: Drug: Aliskiren; Drug: Placebo to aliskiren; Drug: Placebo to valsartan
- Valsartan (Active Comparator): For the first week of the 8 week treatment period, patients received valsartan 160 mg, placebo to valsartan, and 2 tablets of placebo to aliskiren. For the remaining 7 weeks of the study, patients received valsartan 320 mg (two 160 mg capsules) and 2 tablets of placebo to aliskiren. The tablets and capsules (2 of each) were taken orally once daily each morning. To evaluate a missed dose, the last dose of medication was administered at the clinic, and the patient was scheduled to return 2 days later for exercise testing (8 weeks + 2 days).
  Interventions: Drug: Valsartan; Drug: Placebo to aliskiren; Drug: Placebo to valsartan

INTERVENTIONS:
Drug: Aliskiren — Aliskiren was supplied in 150 mg tablets.
  Arms: Aliskiren
Drug: Valsartan — Valsartan was supplied in 160 mg capsules.
  Arms: Valsartan
Drug: Placebo to aliskiren — Placebo to aliskiren was supplied in tablets matching aliskiren 150 mg.
Drug: Placebo to valsartan — Placebo to valsartan was supplied in capsules matching valsartan 160 mg.

SUMMARY:
This study compared the blunting effect of aliskiren and valsartan monotherapies on exercise-induced rises in systolic blood pressure in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion criteria:

* Mean sitting systolic blood pressure ≥ 140 mmHg and < 180 mmHg measured at rest
* Patients able to exercise and to reach 85% of their predicted heart rate during a standard exercise test on a treadmill according to the Bruce Protocol

Exclusion criteria:

* Patients not confident in exercising or not able to exercise
* Absolute contraindication to exercise
* Mean sitting systolic blood pressure ≥ 180 mmHg and/or mean sitting diastolic blood pressure ≥ 110 mmHg measured at rest

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (8):
- Czechia (2):
  - Investigative Site, Pardubice
  - Investigative Site, Prague
- Hungary (4):
  - Investigative Site, Budapest
  - Investigative Site, Nyíregyháza
  - Investigative Site, Pilisvörösvár
  - Investigative Site, Szentendre
- Investigative Site, Singapore, Singapore
- Investigative Site, Leicester, United Kingdom

REFERENCES:
- [Derived] Wang GM, Li LJ, Fan L, Xu M, Tang WL, Wright JM. Renin inhibitors versus angiotensin receptor blockers for primary hypertension. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD012570. doi: 10.1002/14651858.CD012570.pub2. PMID 40013543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients underwent a 2-week washout and a 1-2 week single blind placebo run in. Eligible patients then performed the treadmill exercise test for randomization according to the Bruce Protocol. Patients capable of reaching the defined peak exercise (85% of their predicted HR) were randomized into the study.
Period: Overall Study
Arm/Group | Aliskiren | Valsartan
Started | 33 | 35
Completed | 32 | 33
Not Completed | 1 | 2
Not completed — Unsatisfactory therapeutic effect | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Valsartan | Total
Number analyzed (Participants) | 33 | 35 | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (6.3) | 60 (8.3) | 59 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 19 | 27 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting vs. Peak Heart Rate Systolic Blood Pressure (SBP) From Baseline to Week 8 After a Missed Dose
Description: The difference in resting vs. peak (85% of maximal predicted) heart rate (HR) SBP was calculated by measuring SBP before and during exercise on a standardized treadmill test, conducted according to the Bruce Protocol. Treadmill speed and incline were increased every 3 minutes until the patient was exhausted or peak HR was reached. The SBP at rest vs peak HR was recorded at Baseline and at Week 8 + 2 days (24-hrs after a missed dose); the change in rest vs. peak SBP between these timepoints is reported. The analysis included the rest to peak increase in SBP at baseline as a covariate.
Time Frame: Baseline and Week 8 + 2 days (48-hours after the last dose; 24 hours after a missed dose). Blood Pressure measurements were taken at rest and at peak heart rate at both timepoints.
Population: The Full Analysis Set (FAS) consisted of all patients who were randomized and took at least one dose of study drug. The Exercise Evaluable Set (EES) included all patients included in the FAS for whom the treadmill test values for SBP at peak were available at baseline and after a missed dose.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren | Valsartan
Number analyzed (Participants) | 32 | 33
mmHg | 2.58 (3.54) | 8.26 (3.48)

2. Secondary Outcome: Change in Resting vs. Peak Heart Rate Systolic Blood Pressure (SBP) From Baseline to Week 8
Description: The difference in resting vs. peak (85% of the maximal predicted) heart rate (HR) SBP was calculated by measuring SBP before and during exercise on a standardized treadmill test, conducted according to the Bruce Protocol. Treadmill speed and incline were increased every 3 minutes until the patient was exhausted or peak HR was reached. The SBP at rest vs peak HR was recorded at Baseline and at Week 8 (end of active treatment); the change in SBP between these timepoints is reported. The analysis included the rest to peak increase in SBP at baseline as a covariate.
Time Frame: Baseline and Week 8 (end of active treatment). Blood Pressure measurements were taken at rest and at peak heart rate at both timepoints.
Population: The Full Analysis Set (FAS) consisted of all patients who were randomized and took at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren | Valsartan
Number analyzed (Participants) | 32 | 33
mmHg | 5.78 (3.22) | 7.79 (3.18)

3. Secondary Outcome: Change in Resting vs. Peak Heart Rate Systolic Blood Pressure (SBP) From Week 8 (End of Active Treatment) to 24-hours After a Missed Dose
Description: The difference in resting vs. peak (85% of maximal predicted) heart rate (HR) SBP was calculated by measuring SBP before and during exercise on a standardized treadmill test, conducted according to the Bruce Protocol. The SBP at rest vs peak HR was recorded at Week 8 (end of active treatment) and Week 8 + 2 days (48-hrs after last dose; 24-hrs after missed dose); the change in rest vs. peak SBP between these timepoints is reported. The analysis included the rest to peak increase in SBP at baseline as a covariate.
Time Frame: Week 8 (Last dose; end of active treatment) and Week 8 + 2 days (48-hours after the last dose; 24 hours after a missed dose). Blood Pressure measurements were taken at rest and at peak heart rate at both timepoints.
Population: The Full Analysis Set (FAS) consisted of all patients who were randomized and took at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren | Valsartan
Number analyzed (Participants) | 32 | 33
mmHg | -4.16 (3.28) | 1.37 (3.16)

ADVERSE EVENTS:
Arm/Group | Aliskiren | Valsartan
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 3/33 | 4/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=33) | Valsartan (N=35)
Bronchitis (Infections and infestations) | 0 | 2
Headache (Nervous system disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.